CLINICAL TRIAL: NCT01385982
Title: Improving Management of Outpatient Actionable Test Results
Acronym: OutptATR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Rothschild, MD, Hospitalist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011P000035; 1R18HS019603-01 (AHRQ)
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Management of Actionable Test Results (ATRs)
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Actionable Test Results (Other): Creating standardized policies and procedures around actionable test results (ATR) management, and implementing them network-wide:
  1. Defining the levels of severity and urgency for clinically significant test results
  2. Network-wide policy for test result follow-up by the responsible providers, documentation and escalation processes to assure timely communication.
  3. Standardized policies for the time frames and nature of communication of test result alerts.
  4. Establish criteria for appropriate ATR management by the responsible provider.
  5. Feedback performance including provider, practice and service report cards
  Interventions: Other: Actionable Test Result Management/Standardization

INTERVENTIONS:
Other: Actionable Test Result Management/Standardization — The intervention includes enterprise-wide standardization of actionable test result (ATR) definitions with stratification of significant results into alert levels, expected timeframes for clinician responses, a set of policies for ATR follow-up, metrics to measure ATR management and performance feedback.

SUMMARY:
Clinically significant test results require timely clinician follow-up including the non-urgent clinically significant, or actionable, test results that have received less standardized management and attention. Unfortunately, failure to correctly manage actionable test results is not infrequent and may be associated with important delays in diagnosis and treatment and patient harm. The investigators have designed a safe practice intervention to improve the management of actionable test results for ambulatory patients in a large healthcare system.

ELIGIBILITY:
Inclusion Criteria:

Primary care physicians will be enrolled in the study by virtue of being an actively practicing clinician in an PHS ambulatory practice, and having at least one patient with a diagnostic test included in the PHS CCSTR intervention. The patient population will consist of adult patients >17 years of age with diagnostic tests in the affiliated ambulatory practices of PHS. Patients will be recruited into the study by a review of electronic medical record data to identify patients with a diagnostic test specified in the PHS CCSTR intervention.

Exclusion Criteria:

Participants who do not meet the inclusion/eligibility requirements will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Acknowledged Sub-Critical/Abnormal ATRs | Acknowledgement within 15 business days from the Level 3 Laboratory ATR alert and acknowledgement within 8 business hours of the cardiology Level 2 ATR alert
  The primary outcome of interest is the proportion of sub-critical/abnormal (Level 3 Laboratory and Level 2 Cardiology) ATRs documented as acknowledged by the responsible clinician and having appropriate, follow-up action(s).

SECONDARY OUTCOMES:
Diagnosis and/or Treatment Delays | Minumum of 3 months post ATR
  The frequency of delays to diagnoses and/or treatment of conditions of interest
Undiagnosed/Untreated Condition Frequency and Severity | Minumum of 3 months post ATR
  The frequency and severity of undiagnosed or untreated conditions of interest that occur during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rothschild, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners Healthcare, Boston, Massachusetts, United States